CLINICAL TRIAL: NCT06468176
Title: Efficacy of a Mixed Distancial Neuropsychological Rehabilitation Program in Patients With Grade 2 or 3 Diffuse Glioma : a Randomized Controlled Trial
Brief Title: Efficacy of a Mixed Distancial Neuropsychological Rehabilitation Program in Patients With Grade 2 or 3 Diffuse Glioma
Acronym: FREEDOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROICM 2023-06 FRE
Record Dates: First submitted 2024-05-17; First posted 2024-06-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Glioma, Malignant
Keywords: Oncology; Neurologic Disorder; Neuropsychological rehabilitation; Diffuse Glioma
MeSH Terms: conditions — Glioma; Neoplasms; Nervous System Diseases | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Study therapy will include a mixed intervention by a neuropsychologist and a program based on a digital tool
  Interventions: Other: Cognitive Behavioral Therapy (CBT) neuropsychologist
- Control group (No Intervention): Usual management of the cognitive complaint according to the habits of center

INTERVENTIONS:
Other: Cognitive Behavioral Therapy (CBT) neuropsychologist — * CBT: at least 3 teleconsultations by the neuropsychologist (up to 1/week maximum)
  * Brain Head Quarters (BrainHQ) Digital program: 4 sessions of 40 minutes / week
  Other Names: digital program
  Arms: Intervention group

SUMMARY:
Diffuse low-grade glioma are rare brain tumors affecting young subjects (median age at diagnosis 38 years for grade 2 and 49 years for grade 3). Cognitive symptoms are common in these patients, including memory, attention and executive function disorders. These disorders may have a deleterious impact on patients' professional, family and social lives, and have a negative impact on their quality of life. The benefits of cognitive rehabilitation have been demonstrated in other neurological pathologies. Furthermore, due to limited access to rehabilitation by neuropsychologists, some studies have evaluated the impact of digital cognitive rehabilitation programs. However, it cannot replace human support.

DETAILED DESCRIPTION:
Diffuse Low-Grade Gliomas (DLGG) are rare tumors that affect young subjects (median age at diagnosis 38 years for grade 2 and 49 for grade 3). Overall survival varies from 5 to 15 years. Cognitive symptoms are common in these patients, notably impaired memory, attention and executive functions. For examples, in a prospective study conducted by our team, 40-53% of patients with grade 2 DLGG starting first-line chemotherapy had a cognitive complaint. These findings are in line with a recent meta-analysis based on 11 studies involving 313 glioma patients. These cognitive disorders can have a deleterious impact on patients' professional, family and social lives, and have a negative impact on their quality of life. The value of cognitive rehabilitation has been demonstrated in other neurological pathologies. Randomized controlled trials in DLGG are promising, but are ultimately few in number and/or have significant limitations (e.g. small number of patients, sample heterogeneity, questionable matching criteria, lack of control group). Furthermore, due to limited access to rehabilitation by neuropsychologists, some studies have evaluated the impact of digital cognitive rehabilitation programs. Although this type of tool seems particularly well suited to this young patient population, it cannot replace human accompaniment by a neuropsychologist. Indeed, we know the importance of the patient's human therapeutic alliance for adherence to a program. Moreover, certain psychopathological variables (e.g. anxiety, depression) have a significant impact on both neurocognitive abilities and complaints, justifying the intervention of a neuropsychologist specialized in oncology.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, no age limit;
* Histo-molecular diagnosis of grade 2 or 3 diffuse glioma according to World Health Organization (WHO) Classification 2016, regardless of oncological treatments previously received;
* Patient in satisfactory general condition for the study, defined by a WHO performance index ≤ 2 (ECOG-Performance Status (PS) ≤ 2);
* Neurosurgical excision (excluding biopsy) performed ≥ 12 months previously;
* In the case of oncological treatment, patient who has completed his sessions (radiotherapy, chemotherapy) for ≥ 6 months;
* Patient presenting a cognitive complaint defined as a response rated at least "Fairly" to at least one of the 2 items (n°20 and 25) assessing cognitive complaint in the EORTC QLQ-C30 questionnaire (i.e., defined as a score on the "Cognitive Functioning" scale ≤ 66.67);
* Fluent in French;
* Affiliation to the French Social Security System;
* Possible regular use of a digital tool with Internet access;
* Signature of informed consent prior to any study procedure.

Exclusion Criteria:

* Visual or auditory deficit not corrected to normal and/or preventing use of computer tools (i.e., homonymous lateral hemianopia is not a criterion for non-inclusion) ;
* Concurrent participation in a study with cognition as primary endpoint (e.g., "POLCA", " POLO " clinical trials) ;
* Legal incapacity or physical, psychological, social or geographical conditions preventing the patient from signing the consent form or completing the study ;
* Unstable or uncontrolled psychiatric syndrome (i.e., psychotropic treatments are not a criterion for non-inclusion if doses are stable) ;
* Known severe cognitive impairment (e.g., neurodegenerative disease, sequelae of head trauma, etc.) or defined by a score ≤ 20 on the MoCA test or impacting the ability to use digital tools at home ;
* Oncological treatment (radiotherapy and/or chemotherapy and/or surgery) planned within 4 months of inclusion. Targeted anti-Isocitrate DeHydrogenase (IDH) therapies are authorized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Score in the Perceived Cognitive Impairment (PCI) subscale of Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) questionnaire | 4 months
  The FACT-Cog is a self-assessment questionnaire to estimate memory, attention, concentration, language, and thinking abilities of patients before, during, and after chemotherapy. This questionnaire, composed of 37 items consists of four subscales: cognitive impairments perceived by the patient (20 items), comments from others (4 items), cognitive abilities perceived by the patient (9items), and impact on quality of life (4 items). The Perceived Cognitive Impairments and the Comments from Others subscales are rated on 5-point Likert-type scale (from 0 = "Never" to 4 = "Several times a day"). An intensity 5-point Likert-type scale (from 0 "Not at all" to 4 "Very much") is used to rate perceived cognitive abilities and the impact on quality of life. For all subscales, a higher score represents better cognitive functioning or quality of life

SECONDARY OUTCOMES:
Score in the PCI subscale of FACT-Cog questionnaire | 6, 12 and 18 months
  The FACT-Cog is a self-assessment questionnaire to estimate memory, attention, concentration, language, and thinking abilities of patients before, during, and after chemotherapy. This questionnaire, composed of 37 items consists of four subscales: cognitive impairments perceived by the patient (20 items), comments from others (4 items), cognitive abilities perceived by the patient (9items), and impact on quality of life (4 items). The Perceived Cognitive Impairments and the Comments from Others subscales are rated on 5-point Likert-type scale (from 0 = "Never" to 4 = "Several times a day"). An intensity 5-point Likert-type scale (from 0 "Not at all" to 4 "Very much") is used to rate perceived cognitive abilities and the impact on quality of life. For all subscales, a higher score represents better cognitive functioning or quality of life.
Score in the " Comments from the others " subscale of the FACT-Cog | At baseline, 4, 6, 12 and 18 months
  The FACT-Cog is a self-assessment questionnaire to estimate memory, attention, concentration, language, and thinking abilities of patients before, during, and after chemotherapy. This questionnaire, composed of 37 items consists of four subscales including comments from other (4 items). This subscale is rated on 5-point Likert-type scale (from 0 = "Never" to 4 = "Several times a day"). A higher score represents better cognitive functioning or quality of life.
Score in the " Cognitive abilities perceived by the patient " subscale of the FACT-Cog | At baseline, 4 months, 6 months, 12 months, 18 months
  The FACT-Cog is a self-assessment questionnaire to estimate memory, attention, concentration, language, and thinking abilities of patients before, during, and after chemotherapy. This questionnaire, composed of 37 items consists of four subscales including cognitive abilities perceived by the patient (9 items). An intensity 5-point Likert-type scale (from 0 "Not at all" to 4 "Very much") is used to rate perceived cognitive abilities. A higher score represents better cognitive functioning or quality of life.
Score in the " Impact on quality of life " subscale of the FACT-Cog | At baseline, 4 months, 6 months, 12 months, 18 months
  The FACT-Cog is a self-assessment questionnaire to estimate memory, attention, concentration, language, and thinking abilities of patients before, during, and after chemotherapy. This questionnaire, composed of 37 items consists of four subscales including impact on quality of life (4 items). An intensity 5-point Likert-type scale (from 0 "Not at all" to 4 "Very much") is used to rate the impact on quality of life. A higher score represents better cognitive functioning or quality of life.
FACT-Cog cognitive complaints questionnaire and the main neurocognitive domains | At baseline, 4 months and 12 months
  Correlations between scores on the 4 subscales of the FACT-Cog cognitive complaints questionnaire and the main neurocognitive domains (score on global functioning, executive functions, language, working memory, processing speed and social cognition).
Score in the 2 scales of Prospective and Retrospective Memory Questionnaire (PRMQ) for patient and family caregiver | At baseline, 4 months, 6 months, 12 months, 18 months
  The Prospective and Retrospective Memory Questionnaire (PRMQ) is one of the most commonly used scales to assess both retrospective memory (RM) and prospective memory (PM) complaints. The PRMQ is a 16-item, self-report measure of prospective and retrospective failures in everyday life. 8 items enquire about PM and 8 enquire about RM. The items were also designed to contain an equal number of items concerned with either self-cued memory or environmentally-cued memory, and with short-term versus long-term memory.
Difference in score on psychopathological distress via Hospital Anxiety and Depression Scale (HADS) | At baseline, 4 months, 6 months, 12 months, 18 months
  The HADS is a 14 items questionnaire: 7 items related to anxiety and 7 items related to depression scored on a scale. Scores for items in each subscale of the HADS are summed to produce an anxiety score (HADS-A) or a depression score (HADS-D), or can be added to produce a total score corresponding to emotional distress (HADS-T). Each item is rated on a 4-point Likert scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), for a total score ranging from 0-21 for each subscale. The entire scale (emotional distress) range from 0 to 42, with higher scores indicating more distress
Difference in score on quality of life questionnaire Quality of Life Questionnaire - Core (30EORTC QLQ-C30) | At baseline, 4 months, 6 months, 12 months, 18 months
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials. The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Difference in score on quality of life questionnaire Quality of Life Questionnaire - Brain Neoplasm (EORTC QLQ-BN20) | At baseline, 4 months, 6 months, 12 months, 18 months
  This EORTC brain cancer specific questionnaire is intended to supplement the QLQ-C30. The QLQ-BN20 contains 20 items organized into four scales (three items each: future uncertainty, visual disorder, motor dysfunction, and communication deficit), and seven single items (headaches, seizures, drowsiness, hair loss, itchy skin, weakness of legs, and bladder control). All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale, with higher scores indicating more severe symptoms.
Difference in score on fatigue via Multidimensional Fatigue Inventory (MFI-20) | At baseline, 4 months, 6 months, 12 months, 18 months
  The MFI-20 is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. The patient positions himself on a 5-point scale, according to the fatigue he felt the days before the assessment. The " strongly agree " position is worth 5 points, and the " strongly disagree " position is worth 1 point. The score is calculated by adding up the points on the scale. The higher is the score, the more severe is the the fatigue.
Compliance of intervention | 4 months
  Patient adherence to the intervention defined as completion of at least 25 hours of the digital program out of the recommended 40 hours (calculated automatically by the software), and completion of the 3 neuropsycho-oncology (tele)consultations
Difference in score on neurocognitive test via Montreal Cognitive Assessment (MoCA) | At baseline and 4 and 12 months, respectively
  Lasting 10 to 15 minutes, the test assesses mild to moderate cognitive dysfunction, evaluating the following functions: attention, concentration, executive functions, memory, language, visuo-constructive abilities, abstraction skills, calculation, orientation.
2 scores on the Prospective and Retrospective Memory Questionnaire (PRMQ) and the main cognitive domains | At baseline, 4 months and 12 months
  Correlations between the 2 scores on the PRMQ and the main cognitive domains (score for global functioning, executive functions, language, working memory, processing speed and social cognition)
Proportion of patients returning to work | At baseline, 4 months, 6 months, 12 months, 18 months
  Proportion of patients returning to work or increasing their working hours
Difference in score on depression via Beck Depression Inventory II (BDI-II) | At baseline, 4 months, 6 months, 12 months, 18 months
  The Beck Depression Inventory is used to detect depression and its severity. It is a self-assessment test with 21-items and 4 types of response. These range from 0 to 3 and describe the extent to which we identify the reality described. 0 means not identifying at all and 3 describes a fact which identify almost 100%. Four basic categories are established according to the results obtained : 0-13 = low depression, 14-19 = mild depression, 20-28 = moderate depression and 29-63 = severe depression.
Difference in score on anxiety via State-Trait Anxiety Inventory (STAI-Y) | At baseline, 4 months, 6 months, 12 months, 18 months
  The STAI-Y is a test designed to assess momentary and habitual anxiety. It comprises 2 scales of 20 items each: anxiety-state scale assesses the feelings of apprehension, tension, nervousness and concerns that the subject feels at the time of the consultation. It is an indicator of transient changes in anxiety caused by therapeutic or aversive situations.
  The anxiety-trait scale assesses the feelings of apprehension, tension, nervousness and concerns that the subject usually experiences. The purpose of this scale is to identify anxiety as a stable disposition. It thus forms the starting point for therapeutic action.
  The STAI-Y is also used to study the effect of anxiety on memory, learning performance or adjustment to stressful situations
Difference in score on irritability via Brief Irritability Test (BIT) for patient and family caregiver | At baseline, 4 months, 6 months, 12 months, 18 months
  The Brief Irritability Test is a brief, reliable, and valid self-report measure of irritability with 5-items. The answers are rated from never to always.
Difference in score on insomnia via Insomnia Severity Index (ISI) | At baseline, 4 months, 6 months, 12 months, 18 months
  The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia. The usual recall period is the "last month" and the dimensions evaluated are: severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Difference in score on cognitive abilities index via Wechsler Adult Intelligent Scale (WAIS-IV) | At Baseline, 4 months, 12 months
  This test assesses cognitive abilities across various domains. It comprises 10 core subtests that yield four factor index scores (i.e., Verbal Comprehension: measures language use and long-term memory, Perceptual Reasoning: assesses logical reasoning and visual-spatial abilities, Working Memory: evaluates short-term memory, and Processing Speed: gauges processing speed) as well as the full-scale IQ. There are also five supplemental subtests that can be used as an alternative to the core subtests. In the FREEDOME study, the following sub-tests will be used:
  * Digit Symbol Substitution Test
  * Code test
  * Verbal Digit-span test
  * Arithmetic
Difference in score on verbal learning and memory via Hopkins Verbal Learning Test (HVLT) | At Baseline, 4 months, 12 months
  This test provides a measure of verbal learning and memory. Following each administration, subjects were asked for an immediate free recall. Twenty minutes later, used for intercurrent tasks, subjects were asked for a delayed free recall, which was immediately followed by a recognition memory task. In this task, subjects listened to a list of 24 words, 12 belonging to the studied list and 12 were distractors; the subjects were asked to recognize the 12 studied words.
Difference in score on processing speed and executive function via Stroop Delis-Kaplan test | At Baseline, 4 months, 12 months
  The Delis-Kaplan Executive Function System (D-KEFS) Color-Word-Interference Test (CWIT; AKA Stroop test) is a widely used measure of processing speed and executive function. The Stroop test assesses the interference between color and word reading. Participants are presented with a list of color names (e.g., "red," "blue," "green") printed in incongruent colors (e.g., the word "red" printed in blue ink). The task requires individuals to name the color of the ink while inhibiting the automatic response to read the word itself. The interference effect occurs because our brains process the meaning of the word faster than the color information.
Difference in score on verbal fluency via verbal fluency test | At Baseline, 4 months, 12 months
  Two kinds of verbal fluency (VF) can be differentiated: phonemic fluency refers to the ability to name words with a given first letter (such as "S" or "P"), while in semantic VF words belonging to certain categories such as animals or fruits have to be enumerated. VF is an integral part of many neuropsychological test batteries
Difference in score on visual attention via Trail Making Test (TMT) | At Baseline, 4 months, 12 months
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It comprises two parts in which the subject must connect a set of 25 points as quickly as possible while maintaining accuracy, i.e. avoiding making mistakes. The test provides information on visual search speed, visual exploration, information processing speed, mental flexibility and executive functioning.
Difference in score on Theory of Mind via Reading the Mind in the Eyes Test (RMET) | At Baseline, 4 months, 12 months
  The Reading the Mind in the Eyes Test (RMET) is a common measure of the Theory of Mind.
  In the RMET, participants are presented with pictures of the eye regions of a face and required to select the word that best matches the model's complex mental state such as desire and goal.
  It presents thirty-six photographs of the eye part of the face, each expressing complex mental states of the individuals pictured.

CONTACTS AND LOCATIONS:
Overall Officials: Amelie DARLIX, MD, Study Chair — Institut de Cancérologie de Montpellier (ICM); Estelle GUERDOUX, PHD, Principal Investigator — Institut de Cancérologie de Montpellier (ICM)
Locations (8):
- France (8):
  - Institut régional du Cancer de Montpellier, Montpellier, Hérault
  - CHU Amiens, Amiens
  - CHU Bordeaux, Bordeaux
  - CHU Lyon, Lyon
  - Hôpital de la Timone, Marseille
  - CHU Nancy, Nancy
  - CHU Nîmes, Nîmes
  - Institut Claudius Régaud, Toulouse

REFERENCES:
- [Derived] Guerdoux E, Coutant L, Gourgou S, Mollevi C, Duc MS, Salasc F, Duffau H, Darlix A. Efficacy of hybrid remote neuropsychological rehabilitation on cognitive complaints in post-therapeutic lower-grade glioma: the FREEDOME randomized study protocol. Front Psychol. 2025 Sep 23;16:1650861. doi: 10.3389/fpsyg.2025.1650861. eCollection 2025. PMID 41064168